CLINICAL TRIAL: NCT04542577
Title: Multicenter PMCF Study on the Safety and Performance of PROSPACE 3D / PROSPACE 3D OBLIQUE / TSPACE 3D - A Prospective Study on Total Indications
Brief Title: PMCF Study on the Safety and Performance of PROSPACE 3D / PROSPACE 3D OBLIQUE / TSPACE 3D
Acronym: PROTONTO
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2003
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Degenerative Instability; Spondylolisthesis; Post-discectomy Syndrome; Post-traumatic Instabilities
Keywords: Lumbar interbody Fusion; Intervertebral Implant
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, pure data collection of all PROSPACE 3D, PROSPACE 3D Oblique, TSPACE 3D patients in selected centers (not interventional, multicenter

DETAILED DESCRIPTION:
The study collects a data set for each patient receiving a PROSPACE 3D, PROSPACE 3D Oblique, or TSPACE 3D implant. It is intended to collect data preoperatively, intraoperatively and at one follow-up- assessment after a minimum of one year postoperatively containing

* Basic medical history
* Type of surgical procedure
* Treated segments
* Implant characteristics (including additional implants for anterior/posterior stabilization)
* Scores: ODI, Pain (VAS), EQ-5D
* Patient satisfaction

ELIGIBILITY:
Inclusion:

* Patient is minimum 18 years old
* Written informed consent for the documentation of clinical and radiological results
* Patient's indication according to IFU
* Patient is not pregnant

Exclusion:

- Patient is not willing or able to participate at the follow-up examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients undergoing PROSPACE 3D, PROSPACE 3D OBLIQUE or TSPACE 3D surgery in the participating Hospitals meeting the inclusion criteria are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Change of Spinal Disability measured by Oswestry Disability Index (ODI) | preoperatively, at 3 months postoperatively and at 12 months postoperatively
  The Oswestry Disability Index (ODI) is designed to measure back-specific disability. The questionnaire has 10 items concerning pain and activities of daily living including pain, personal care, lifting, Walking, sitting, standing, sleeping, sex life, social life and travelling. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

SECONDARY OUTCOMES:
Change of Pain (VAS) | preoperatively, at 3 months postoperatively and at 12 months postoperatively
  Pain will be assessed by the patient using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal/worst pain"
Change of Quality of Life (EQ-5D) | preoperatively, at 3 months postoperatively and at 12 months postoperatively
  The score is self-completion by the patient and will therefore be used in German. The Quality of Life Score "EQ-5D" is a standardized 5-dimension 5-level measure of the health status and is developed by the EuroQol Group in order to have a simple and generic measure for clinical and economic assessment. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Bone fusion | 12 Months postoperatively
  After IBF surgery fusion of the treated segment is aspired. Thus, the implant design shall allow on-/ingrowth to/into the material. The fusion status can be determined from radiographs (static or dynamic). Bony fusion can be characterized quantitatively by the fusion rate.
Side effects | up to 12 months postoperatively
  Occurrence of complications potentially associated with the implanted devices can never be fully excluded during spinal surgery. In order to monitor potential complication and to identify so far unknown complications AEs and SAEs deemed related to the investigational device are recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Katholisches Klinikum Koblenz, Koblenz
  - Sana Kliniken Sommerfeld, Kremmen